CLINICAL TRIAL: NCT03028493
Title: Increasing the Accessibility of a Falls Prevention Intervention for Community Dwelling Older Adults With Low Vision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Blaylock (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Sarah Blaylock, Doctoral Candidate Department of Occupational Therapy, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 01633
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Low Vision; Fall
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Three individuals not involved in intervention delivery will complete pre-post measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted SAFE Intervention (Experimental): Adapted version of the SAFE Health Behavior and Exercise intervention.
  Interventions: Behavioral: Adapted SAFE Intervention
- Original SAFE Intervention (Active Comparator): Original version of the SAFE intervention.
  Interventions: Behavioral: Original SAFE Intervention

INTERVENTIONS:
Behavioral: Original SAFE Intervention — A CDC recommended, evidence-based falls prevention intervention.
  Arms: Original SAFE Intervention
Behavioral: Adapted SAFE Intervention — An adapted version of the SAFE intervention meant to target older adults with low vision.
  Arms: Adapted SAFE Intervention

SUMMARY:
This study serves to test a previously evaluated falls prevention intervention recommended by the Centers for Disease Control and Prevention, entitled the Study of Accidental Falls in the Elderly (SAFE) Health Behavior and Exercise Intervention, to evaluate if the intervention is accessible to older adults with low vision receiving services from the Southeastern Blind Rehabilitation Center (SBRC). This study also serves to pilot a version of the SAFE intervention that has been adapted to be accessible for individuals with low vision at SBRC.

DETAILED DESCRIPTION:
This study serves to compare the comprehension and retention of individuals completing a version of the SAFE falls prevention intervention adapted for low vision versus individuals receiving the original intervention. One group of participants will complete the standard SAFE intervention format while another group will complete the same intervention with written materials adapted for those with vision loss. One intervention (either standard or adapted SAFE program) will be delivered at a time. The SAFE intervention is comprised of four, 90-minute group classes that address environmental, behavioral, and physical falls risk factors. Classes involve lecture and group discussions as well as review of low intensity exercises. The adapted content is presented in large print with high contrast and has been rewritten on a lower grade level. A nutritionist, a physical therapist, a physician, 5 older adults with low vision, 10 low vision occupational therapist, and 5 health literacy experts provided feedback to strengthen the adapted intervention.

ELIGIBILITY:
Inclusion Criteria:

* 60 and older;
* Visual impairment with some remaining reading ability.

Exclusion Criteria:

* Less than age 60;
* Complete blindness;
* Vertebral osteoporosis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Change in knowledge of falls prevention | Pre and post (2 weeks after start of intervention delivery)
  10 multiple choice questions based on the SAFE intervention content

SECONDARY OUTCOMES:
Short Physical Performance Battery | Pre
  Measures of balance, gait, and sit to stand
PROMIS Depression Scale | Pre
  Measures depression
PROMIS Participation Scale | Pre
  Measures daily participation
PROMIS Global Health | Pre
  Measures general health
UAB Life-Space Inventory | Pre
  Measures places travelled within past month

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Brown, MD, MSPH, Principal Investigator — Birmingham VA and UAB School of Medicine
Locations (1):
- Department of Veteran Affairs, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
All data serves to fulfill dissertation requirement and will not be shared with additional researchers.